CLINICAL TRIAL: NCT05727098
Title: Comparative Study Between Dexmedetomedine and Ketamine in Erector Spinae Plane Block for Postoperative Analgesia Following Modified Radical Mastectomy. A Prospective Randomized Controlled Study.
Brief Title: Dexmedetomedine and Ketamine in Erector Spinae Block for Postoperative Analgesia Following Mastectomy.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Ehab Hanafy Shaker, Associate Professor of Anesthesia, ICU and Pain management, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Erector block after mastectomy
Record Dates: First submitted 2023-02-03; First posted 2023-02-14 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bupivacaine; Anesthetics, Local; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bupivacaine (Active Comparator): Will receive ultrasound guided ESPB with 0,25% Bupivacaine .
  Interventions: Drug: Bupivacaine Hydrochloride
- Bupivacaine and dexmedetomedine (Active Comparator): Will receive ultrasound guided ESPB with 0,25% Bupivacaine + Dexmedetomidine.
  Interventions: Drug: Bupivacaine Hydrochloride and dexmedetomedine
- Bupivacaine and Ketamine (Active Comparator): will receive ultrasound guided ESPB with 0,25% Bupivacaine + Ketamine.
  Interventions: Drug: Bupivacaine Hydrochloride and ketamine

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride — injection of Bupivacaine 0.25% in ESPB
  Other Names: local anesthetic
  Arms: Bupivacaine
Drug: Bupivacaine Hydrochloride and dexmedetomedine — injection of Bupivacaine 0.25% and dexmedetomedine in ESPB
  Other Names: local anesthetic and dexmedetomedine
  Arms: Bupivacaine and dexmedetomedine
Drug: Bupivacaine Hydrochloride and ketamine — injection of Bupivacaine 0.25% and ketamine in ESPB
  Other Names: local anesthetic and ketamine
  Arms: Bupivacaine and Ketamine

SUMMARY:
Persistent pain after breast cancer surgery is frequently observed in more than 60% of patients.The suboptimal management of perioperative pain can lead to the occurrence of persistent breast cancer pain syndrome and phantom breast pain. Dexmedetomidine, a novel α2-agonist with an eight-fold affinity for α2-adrenergic receptors (sedate and analgesic effects) as clonidine, while exerts much less α1-effects., has been found to significantly increase the duration of peripheral nerve blocks, with minimal systemic side effects.

Ketamine is a non-competitive antagonist of the N-methyl-D-aspartate (NMDA) receptors. It is used for sedation, premedication, induction, and maintenance of general anesthesia. Central, regional, and local anesthetic and analgesic properties have been reported for ketamine. Both can be used through Erector spinae plane block for postoperative pain control.

DETAILED DESCRIPTION:
Persistent pain after breast cancer surgery is frequently observed in more than 60% of patients.The suboptimal management of perioperative pain can lead to the occurrence of persistent breast cancer pain syndrome and phantom breast pain.

A systematic review and meta-analysis of experimental studies showed that the provision of effective analgesia reduces both the number and incidence of metastases in experimental cancer models . Pain may influence body homeostasis and cancer progression by pain-related immune suppression.

General anesthesia is the conventional, most frequently used anesthetic technique in breast cancer surgical interventions. Various regional anesthetic techniques have also been used; these include local wound infiltration, thoracic epidural anesthesia, paravertebral block (PVB), thoracic spinal anesthesia, and more recently, ultrasound-guided interfacial plane blocks such as pectoral nerve (PECS) blocks type 1 and 2 and the serratus plane block (SPB). Recently introduced erector spinae plane block (ESPB) requires less technical expertise (easy), and may be a safe alternative to PVB. ESP block is described for treating thoracic neuropathic pain with encouraging results. ESP is a potential space deep to erector spinae muscle (ES), where the injected local anaesthetic (LA) spreads cranio-caudally up to several levels as the ES fascia extends from nuchal fascia cranially to the sacrum caudally (C7-T2 cranially and L2-L3 caudally), The block covers somatic and visceral pain during breast surgery blocks by blocking ventral rami, dorsal rami of spinal nerves, and rami communicans that transmit sympathetic fibers.

There is another potentially beneficial effects of regional anaesthesia and analgesia on perioperative outcomes, these include decreased opioids consumption , lower rate of post-operative pulmonary complications, decreased post-operative nausea vomiting (PONV) and decreased duration of post-anaesthesia care unit stay. Regional anaesthesia has long-term oncological outcomes as it is considered protective for cancer recurrence by its indirect and direct antiproliferative effects.

Over recent years, the addition of multiple types of additives to local anesthetics has been reported to improve analgesic effect of peripheral nerve block and regional blocks Dexmedetomidine, a novel α2-agonist with an eight-fold affinity for α2-adrenergic receptors (sedate and analgesic effects) as clonidine, while exerts much less α1-effects., has been found to significantly increase the duration of peripheral nerve blocks, with minimal systemic side effects.

Ketamine is a non-competitive antagonist of the N-methyl-D-aspartate (NMDA) receptors. It is used for sedation, premedication, induction, and maintenance of general anesthesia. Central, regional, and local anesthetic and analgesic properties have been reported for ketamine.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II .
* female aged between 18 to 65. Scheduled for elective modified radical mastectomy under general anesthesia.

Exclusion Criteria:

* Patient known to have allergy to any of the drugs used in the study.
* Infection at injection site.
* Coagulation disorders.
* severe heart ,liver or kidney disease.
* Unwillingness.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — gender identity only females
Enrollment: 75 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Time to first rescue analgesia request postoperative | 24 hours
  the time of first rescue analgesia
Total opioid consumption | 24 hours
  Total opioid consumption

SECONDARY OUTCOMES:
Visual analogue scale. | 24 hours
  Calculation of Visual analogue scale at rest and mouvement. It is 10 points scale from 0 to 10 where 0 represents no pain while 10 represents maximum pain

CONTACTS AND LOCATIONS:
Overall Officials: Ehab H Shaker, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Hanafy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
After data publication upon request

REFERENCES:
- [Result] Hasoon J, Urits I, Viswanath O, Dar B, Kaye AD. Erector Spinae Plane Block for the Treatment of Post Mastectomy Pain Syndrome. Cureus. 2021 Jan 12;13(1):e12656. doi: 10.7759/cureus.12656. PMID 33585141
- See also: Erector Spinae Plane Block for the Treatment of Post Mastectomy Pain Syndrome — https://pubmed.ncbi.nlm.nih.gov/33585141/